CLINICAL TRIAL: NCT06721871
Title: Evaluation of Safety, Tolerability and Efficacy of Crofelemer Following Multiple Ascending Doses of Crofelemer Powder for Oral Solution in Pediatric Participants With Microvillus Inclusion Disease (MVID)
Brief Title: Ascending Doses of Crofelemer Powder for Oral Solution in Pediatric Microvillus Inclusion Disease (MVID)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Napo Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NP303-104
Record Dates: First submitted 2024-11-20; First posted 2024-12-06 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Microvillus Inclusion Disease; Congenital Disorders; Rare Diseases
MeSH Terms: conditions — Microvillus inclusion disease; Congenital, Hereditary, and Neonatal Diseases and Abnormalities; Rare Diseases | interventions — Solutions

STUDY DESIGN:
Intervention Model Description: Each dose level will include 2 4-week Treatment Periods for a total of 8 weeks. There will be 3 ascending dose levels for a total of 24 weeks of treatment with either crofelemer or placebo, with safety reviews between dose levels. Within the 24 weeks of treatment, each of crofelemer and placebo will have been administered at 3 ascending dose levels for 4 weeks each, totaling 12 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a randomized, double-blind, placebo-controlled, dose-escalating study with a placebo cross-over design within each participant at each dose level in this ultra-rare MVID participant population
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Dose Level 1/Treatment Period 1: 1mg/kg/dose 3x/day (Experimental): Participants may be randomized to crofelemer powder for oral solution during Treatment Period 1 (1 month duration)
  Interventions: Drug: Crofelemer Powder for Oral Solution
- Dose Level 1/Treatment Period 1: Placebo 3x/day (Placebo Comparator): Participants may be randomized to the placebo comparator during Treatment Period 1 (1 month duration)
  Interventions: Drug: Placebo Powder for Oral Solution
- Dose Level 1/Treatment Period 2: 1mg/kg/dose 3x/day (Experimental): Participants will crossover to either crofelemer powder for oral solution or placebo comparator
  Interventions: Drug: Crofelemer Powder for Oral Solution
- Dose Level 2/Treatment Period 1: 3mg/kg/dose 3x/day (Experimental): Participants will crossover to either crofelemer powder for oral solution or placebo comparator or continue on crofelemer powder for oral solution or the placebo comparator that they were previously on during Dose Level 1 (1 month duration)
  Interventions: Drug: Crofelemer Powder for Oral Solution
- Dose Level 2/Treatment Period 1: Placebo 3x/day (Placebo Comparator): Participants will crossover to either crofelemer powder for oral solution or placebo comparator or continue on crofelemer powder for oral solution or the placebo comparator that they were previously on during Dose Level 1 (1 month duration)
  Interventions: Drug: Placebo Powder for Oral Solution
- Dose Level 2/Treatment Period 2: 3mg/kg/dose 3x/day (Experimental): Participants will crossover to either crofelemer powder for oral solution or placebo comparator
  Interventions: Drug: Crofelemer Powder for Oral Solution
- Dose Level 2/Treatment Period 2: Placebo 3x/day (Placebo Comparator): Participants will crossover to either crofelemer powder for oral solution or placebo comparator
  Interventions: Drug: Placebo Powder for Oral Solution
- Dose Level 3/Treatment Period 1: 10mg/kg/dose 3x/day (Experimental): Participants will crossover to either crofelemer powder for oral solution or placebo comparator or continue on crofelemer powder for oral solution or the placebo comparator that they were previously on during Dose Level 2 (1 month duration)
  Interventions: Drug: Crofelemer Powder for Oral Solution
- Dose Level 3/Treatment Period 1: Placebo 3x/day (Placebo Comparator): Participants will crossover to either crofelemer powder for oral solution or placebo comparator or continue on crofelemer powder for oral solutionor the placebo comparator that they were previously on during Dose Level 2 (1 month duration)
  Interventions: Drug: Placebo Powder for Oral Solution
- Dose Level 3/Treatment Period 2: 10mg/kg/dose 3x/day (Experimental): Participants will crossover to either crofelemer powder for oral solution or placebo comparator
  Interventions: Drug: Crofelemer Powder for Oral Solution
- Dose Level 3/Treatment Period 2: Placebo 3x/day (Placebo Comparator): Participants will crossover to either crofelemer powder for oral solution or placebo comparator
  Interventions: Drug: Placebo Powder for Oral Solution
- Dose Level 1/Treatment Period 2: Placebo 3x/day (Placebo Comparator): Participants will crossover to either crofelemer powder for oral solution or placebo comparator
  Interventions: Drug: Placebo Powder for Oral Solution

INTERVENTIONS:
Drug: Crofelemer Powder for Oral Solution — Crofelemer Powder for Oral Solution
  Arms: Dose Level 1/Treatment Period 1: 1mg/kg/dose 3x/day; Dose Level 1/Treatment Period 2: 1mg/kg/dose 3x/day; Dose Level 2/Treatment Period 1: 3mg/kg/dose 3x/day; Dose Level 2/Treatment Period 2: 3mg/kg/dose 3x/day; Dose Level 3/Treatment Period 1: 10mg/kg/dose 3x/day; Dose Level 3/Treatment Period 2: 10mg/kg/dose 3x/day
Drug: Placebo Powder for Oral Solution — Matching Placebo Powder for Oral Solution
  Arms: Dose Level 1/Treatment Period 1: Placebo 3x/day; Dose Level 1/Treatment Period 2: Placebo 3x/day; Dose Level 2/Treatment Period 1: Placebo 3x/day; Dose Level 2/Treatment Period 2: Placebo 3x/day; Dose Level 3/Treatment Period 1: Placebo 3x/day; Dose Level 3/Treatment Period 2: Placebo 3x/day

SUMMARY:
a 32-week study that will evaluate the safety, tolerability and preliminary efficacy of multiple ascending doses of crofelemer, compared to placebo, using a randomized cross-over design within each dose level, when administered to participants with MVID receiving parenteral support (PS, defined as TPN with or without supplementary IV fluid requirements). Blinded study drug will be administered as a novel crofelemer formulation, Crofelemer Powder for Oral Solution, or a matching placebo powder formulation for oral solution. Assigned study drug will be reconstituted and administered orally (or enterally) three times daily (TID) as a concentrated liquid formulation in each of the three dose levels

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, dose-escalating study with a placebo cross-over design within each dose level in this ultra-rare MVID participant population. For the primary objective, safety and tolerability, comparisons between the crofelemer and placebo within each dose level and over 24 weeks with all 3 dose levels combined will be descriptively summarized. For secondary objectives, changes from the 8-week pre-treatment Baseline Period will be made: 1) within each participant between crofelemer and placebo within each dose level, 2) within each participant between crofelemer and placebo through 24 weeks, 3) between the crofelemer and placebo groups (if multiple participants per group are enrolled) within each dose level, and 4) between the crofelemer and placebo groups (if multiple participants per group are enrolled) through 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Participants (assent for participants older than 7 years of age) and/or their legal parent/guardian sign an Informed Consent Form (ICF) indicating that they understand the purpose of the procedures required for the study and are willing to participate
2. When appropriate, pediatric participants, whose age, cognitive skills, reading abilities and maturity allow the understanding of the study protocol should provide written assent to participate.
3. Male or female participants between the ages of 3 months to 17 years at the time of signing the informed consent or providing assent
4. Have a confirmed diagnosis (genetic and/or histologic) of MVID
5. Are able to ingest reconstituted Crofelemer Powder for Oral Solution either orally (PO) or through a previously-placed G-tube or GJ-Tube (not via J-Tube)
6. Have, during the 8 weeks prior to baseline, a volume of PS that represents at least 50% (≥ 50%) of the participant's weekly hydration volume requirements
7. If female participants have reached menarche, the participant (and caregiver) agree that the participant will remain abstinent or use two accepted methods of birth control during the course of the treatment period and for an additional 30 days following the last dose of study drug.
8. Male participants (and caregiver) agree that the participant will remain abstinent or use contraception during the course of the treatment period and continue on for an additional 90 days following the last dose of study drug.

Exclusion Criteria:

Within the last 4 weeks before study initiation, participants have:

1. had significant changes to PS requirements (i.e., ± > 20%)
2. had a new requirement for diuretics
3. had any infection requiring IV antibiotic administration
4. had a documented active gastrointestinal infection
5. initiated any new anti-diarrheal drug
6. had an increase in ALT, AST, or total bilirubin that is ≥2 times the participant's usual laboratory values
7. previously received an organ transplant
8. any currently-diagnosed malignancy
9. is pregnant or breastfeeding
10. any investigator determined criteria for inability to participate in this study

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | 32 Weeks
  Incidence of Adverse Events and Serious Adverse Events
Changes in Physical Examination | 32 Weeks
  Changes from baseline in physical exam and signs of dehydration, such as decreased urine output, sunken eyes, lethargy and abnormal skin turgor.
Changes in laboratory Values | 32 Weeks
  Incidence in changes from baseline of individual lab values within a chemistry, hematology and metabolic panel analysis.

SECONDARY OUTCOMES:
Average Daily Loose/Watery Stool Volume | Average Weekly for 32 weeks
  Measure and record the volume of loose/watery stools each day using a toilet hat for stool collection
Average Daily Stool Frequency | Average Weekly for 32 weeks
  Record the number of stools/day using the Daily Stool Diary
Average Daily Stool Consistency | Average Weekly for 32 weeks
  Record stool consistency of each stool using the 7-point pediatric version of the Bristol Stool Form Scale in the Daily Stool Diary
Stool Electrolyte | Average Weekly for 32 weeks
  Stool electrolyte (Na+, K+, Cl-) concentration measured in mEq/L
PS Volume Requirements | Average Weekly for 32 weeks
  Record daily weekly TPN and IV fluid volume requirements in the Daily TPN and IV Fluid Diary
Average Weekly Supplemental Electrolytes | Average Weekly for 32 Weeks
  Record daily any IV supplements of Na+, K+, Cl-, or acetate on the Daily PS Diary

CONTACTS AND LOCATIONS:
Overall Officials: Lissette Jimenez, MD, MPH, Principal Investigator — Boston Children's Hospital; Pravin Chaturvedi, PhD, Study Chair — Napo Pharmaceuticals, Inc.
Locations (3):
- Boston Children's Hospital, Boston, Massachusetts, United States
- UOS Gastroenterolgia e Riabilitazione nutrizionale Piazza Sant' Onofrio 4, Rome, Italy
- Al Jalila Children's Hospital, Dubai, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Babcock SJ, Flores-Marin D, Thiagarajah JR. The genetics of monogenic intestinal epithelial disorders. Hum Genet. 2023 May;142(5):613-654. doi: 10.1007/s00439-022-02501-5. Epub 2022 Nov 23. PMID 36422736
- [Background] Canani RB, Castaldo G, Bacchetta R, Martin MG, Goulet O. Congenital diarrhoeal disorders: advances in this evolving web of inherited enteropathies. Nat Rev Gastroenterol Hepatol. 2015 May;12(5):293-302. doi: 10.1038/nrgastro.2015.44. Epub 2015 Mar 17. PMID 25782092
- [Background] Berni Canani R, Terrin G, Cardillo G, Tomaiuolo R, Castaldo G. Congenital diarrheal disorders: improved understanding of gene defects is leading to advances in intestinal physiology and clinical management. J Pediatr Gastroenterol Nutr. 2010 Apr;50(4):360-6. doi: 10.1097/MPG.0b013e3181d135ef. PMID 20216094
- [Background] Bowman DM, Kaji I, Goldenring JR. Altered MYO5B Function Underlies Microvillus Inclusion Disease: Opportunities for Intervention at a Cellular Level. Cell Mol Gastroenterol Hepatol. 2022;14(3):553-565. doi: 10.1016/j.jcmgh.2022.04.015. Epub 2022 Jun 1. PMID 35660026
- [Background] Gao JJ, Tan M, Pohlmann PR, Swain SM. HALT-D: A Phase II Evaluation of Crofelemer for the Prevention and Prophylaxis of Diarrhea in Patients With Breast Cancer on Pertuzumab-Based Regimens. Clin Breast Cancer. 2017 Feb;17(1):76-78. doi: 10.1016/j.clbc.2016.08.005. Epub 2016 Aug 27. PMID 27692565
- [Background] Greene C, Barlesi B, Tarroza-David S, Friedlander T. Improved Control of Tyrosine Kinase Inhibitor-Induced Diarrhea with a Novel Chloride Channel Modulator: A Case Report. Oncol Ther. 2021 Jun;9(1):247-253. doi: 10.1007/s40487-021-00147-3. Epub 2021 Apr 7. PMID 33826111
- [Background] Groisman GM, Amar M, Livne E. CD10: a valuable tool for the light microscopic diagnosis of microvillous inclusion disease (familial microvillous atrophy). Am J Surg Pathol. 2002 Jul;26(7):902-7. doi: 10.1097/00000478-200207000-00008. PMID 12131157
- [Background] Hasosah M, Lemberg DA, Skarsgard E, Schreiber R. Congenital short bowel syndrome: a case report and review of the literature. Can J Gastroenterol. 2008 Jan;22(1):71-4. doi: 10.1155/2008/590143. PMID 18209785
- [Background] Knowles BC, Roland JT, Krishnan M, Tyska MJ, Lapierre LA, Dickman PS, Goldenring JR, Shub MD. Myosin Vb uncoupling from RAB8A and RAB11A elicits microvillus inclusion disease. J Clin Invest. 2014 Jul;124(7):2947-62. doi: 10.1172/JCI71651. Epub 2014 Jun 2. PMID 24892806
- [Background] Chowdhury AI, Phillips JF. Predicting contraceptive use in Bangladesh: a logistic regression analysis. J Biosoc Sci. 1989 Apr;21(2):161-8. doi: 10.1017/s0021932000017855. PMID 2722912
- [Background] Leng C, Rings EHHM, de Wildt SN, van IJzendoorn SCD. Pharmacological and Parenteral Nutrition-Based Interventions in Microvillus Inclusion Disease. J Clin Med. 2020 Dec 23;10(1):22. doi: 10.3390/jcm10010022. PMID 33374831
- [Background] Macarthur RD, Hawkins TN, Brown SJ, Lamarca A, Clay PG, Barrett AC, Bortey E, Paterson C, Golden PL, Forbes WP. Efficacy and safety of crofelemer for noninfectious diarrhea in HIV-seropositive individuals (ADVENT trial): a randomized, double-blind, placebo-controlled, two-stage study. HIV Clin Trials. 2013 Nov-Dec;14(6):261-73. doi: 10.1310/hct1406-261. PMID 24334179
- [Background] Mangel AW, Chaturvedi P. Evaluation of crofelemer in the treatment of diarrhea-predominant irritable bowel syndrome patients. Digestion. 2008;78(4):180-6. doi: 10.1159/000185719. Epub 2008 Dec 18. PMID 19092244
- [Background] Muller T, Hess MW, Schiefermeier N, Pfaller K, Ebner HL, Heinz-Erian P, Ponstingl H, Partsch J, Rollinghoff B, Kohler H, Berger T, Lenhartz H, Schlenck B, Houwen RJ, Taylor CJ, Zoller H, Lechner S, Goulet O, Utermann G, Ruemmele FM, Huber LA, Janecke AR. MYO5B mutations cause microvillus inclusion disease and disrupt epithelial cell polarity. Nat Genet. 2008 Oct;40(10):1163-5. doi: 10.1038/ng.225. Epub 2008 Aug 24. PMID 18724368
- [Background] Nee J, Salley K, Ludwig AG, Sommers T, Ballou S, Takazawa E, Duehren S, Singh P, Iturrino J, Katon J, Lee HN, Rangan V, Lembo AJ. Randomized Clinical Trial: Crofelemer Treatment in Women With Diarrhea-Predominant Irritable Bowel Syndrome. Clin Transl Gastroenterol. 2019 Dec;10(12):e00110. doi: 10.14309/ctg.0000000000000110. PMID 31800542
- [Background] Overeem AW, Posovszky C, Rings EH, Giepmans BN, van IJzendoorn SC. The role of enterocyte defects in the pathogenesis of congenital diarrheal disorders. Dis Model Mech. 2016 Jan;9(1):1-12. doi: 10.1242/dmm.022269. PMID 26747865
- [Background] Patel TS, Crutchley RD, Tucker AM, Cottreau J, Garey KW. Crofelemer for the treatment of chronic diarrhea in patients living with HIV/AIDS. HIV AIDS (Auckl). 2013 Jul 15;5:153-62. doi: 10.2147/HIV.S30948. Print 2013. PMID 23888120
- [Background] Phillips AD, Szafranski M, Man LY, Wall WJ. Periodic acid-Schiff staining abnormality in microvillous atrophy: photometric and ultrastructural studies. J Pediatr Gastroenterol Nutr. 2000 Jan;30(1):34-42. doi: 10.1097/00005176-200001000-00015. PMID 10630437
- [Background] Pohlmann PR, Graham D, Wu T, Ottaviano Y, Mohebtash M, Kurian S, McNamara D, Lynce F, Warren R, Dilawari A, Rao S, Mainor C, Swanson N, Tan M, Isaacs C, Swain SM. HALT-D: a randomized open-label phase II study of crofelemer for the prevention of chemotherapy-induced diarrhea in patients with HER2-positive breast cancer receiving trastuzumab, pertuzumab, and a taxane. Breast Cancer Res Treat. 2022 Dec;196(3):571-581. doi: 10.1007/s10549-022-06743-9. Epub 2022 Oct 25. PMID 36280642
- [Background] Ruemmele FM, Schmitz J, Goulet O. Microvillous inclusion disease (microvillous atrophy). Orphanet J Rare Dis. 2006 Jun 26;1:22. doi: 10.1186/1750-1172-1-22. PMID 16800870
- [Background] Terrin G, Tomaiuolo R, Passariello A, Elce A, Amato F, Di Costanzo M, Castaldo G, Canani RB. Congenital diarrheal disorders: an updated diagnostic approach. Int J Mol Sci. 2012;13(4):4168-4185. doi: 10.3390/ijms13044168. Epub 2012 Mar 29. PMID 22605972
- [Background] Thiagarajah JR, Verkman AS. Chloride channel-targeted therapy for secretory diarrheas. Curr Opin Pharmacol. 2013 Dec;13(6):888-94. doi: 10.1016/j.coph.2013.08.005. Epub 2013 Aug 27. PMID 23992767
- [Background] Tradtrantip L, Namkung W, Verkman AS. Crofelemer, an antisecretory antidiarrheal proanthocyanidin oligomer extracted from Croton lechleri, targets two distinct intestinal chloride channels. Mol Pharmacol. 2010 Jan;77(1):69-78. doi: 10.1124/mol.109.061051. Epub 2009 Oct 6. PMID 19808995
- [Background] van der Velde KJ, Dhekne HS, Swertz MA, Sirigu S, Ropars V, Vinke PC, Rengaw T, van den Akker PC, Rings EH, Houdusse A, van Ijzendoorn SC. An overview and online registry of microvillus inclusion disease patients and their MYO5B mutations. Hum Mutat. 2013 Dec;34(12):1597-605. doi: 10.1002/humu.22440. Epub 2013 Oct 16. PMID 24014347
- [Background] Weale AR, Edwards AG, Bailey M, Lear PA. Intestinal adaptation after massive intestinal resection. Postgrad Med J. 2005 Mar;81(953):178-84. doi: 10.1136/pgmj.2004.023846. PMID 15749794
- [Background] Wiegerinck CL, Janecke AR, Schneeberger K, Vogel GF, van Haaften-Visser DY, Escher JC, Adam R, Thoni CE, Pfaller K, Jordan AJ, Weis CA, Nijman IJ, Monroe GR, van Hasselt PM, Cutz E, Klumperman J, Clevers H, Nieuwenhuis EE, Houwen RH, van Haaften G, Hess MW, Huber LA, Stapelbroek JM, Muller T, Middendorp S. Loss of syntaxin 3 causes variant microvillus inclusion disease. Gastroenterology. 2014 Jul;147(1):65-68.e10. doi: 10.1053/j.gastro.2014.04.002. Epub 2014 Apr 12. PMID 24726755